CLINICAL TRIAL: NCT02002013
Title: The Fluid Translation of Research Into Practice Study (Fluid-TRIPS): An International Cross-Sectional Survey of Fluid Resuscitation Practice
Brief Title: The Fluid Translation of Research Into Practice Study
Acronym: Fluid-TRIPS
Status: Completed | Type: Observational
Sponsor: The George Institute for Global Health, Australia (Other)
Responsible Party: Principal Investigator, Naomi Hammond, Co-principle investigator, The George Institute for Global Health, Australia
Other Study IDs: GI-CCT300413; ACTRN12613001172796 (Other: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Critical Care, Fluid Resuscitation
Keywords: Adult; ICU patient; Fluid resuscitation; observational study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult ICU patient receiving Fluid resus: Adult patients present in the ICU at the start of the study day or admitted during the 24-hour study period will be included in the study sample.

SUMMARY:
Translating reliable evidence on fluid resuscitation of intensive care patients into clinical practice - Improving patient outcomes and containing public health costs

DETAILED DESCRIPTION:
The Fluid-Translation of Research into Practice Study (TRIPS) is an international, single day, cross-sectional study planned for the second quarter of 2014, coordinated by the George Institute for Global Health, with the purpose of documenting prescribing practices for fluid resuscitation in intensive care units (ICUs) worldwide. This international cross-sectional study follows on from the publication of large-scale randomized controlled trials and meta-analyses of fluid resuscitation, which provide evidence of how fluid resuscitation may affect patient-centered outcomes.

Fluid-TRIPS is a repeat of the Saline versus Albumin for Fluid Evaluation (SAFE)-TRIPS which was an international cross-sectional survey conducted in 2007 that had 391 ICU's participate from 25 countries and provided insight into international fluid resuscitation practice at that time. Along with establishing if fluid resuscitation practices have changed since SAFE-TRIPS, Fluid-TRIPS also aims to determine the relationship between fluid choice and evidence, along with understand other factors that may influence the choice of bolus fluid in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Adult patients present in the ICU on the study day or admitted during the 24-hour study period will be included in the study sample.

Exclusion Criteria:

Children under 16 years are excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients present in the ICU on the study day
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Type of resuscitation fluid in ICU | 24-hour study day
  To describe the amount and type of resuscitation fluid currently administered to adult patients in intensive care units (ICU) in different countries

SECONDARY OUTCOMES:
Cost comparison of fluid choice between regions | Designated 24-hour study day
  To describe and compare the costs of fluid choice between different geographical regions

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hammond, Study Chair — The George Institute; Colman Taylor, Study Chair — The George Institute
Locations (1):
- The The George Institute for global health; Critical Care & Trauma Division, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Hammond NE, Taylor C, Finfer S, Machado FR, An Y, Billot L, Bloos F, Bozza F, Cavalcanti AB, Correa M, Du B, Hjortrup PB, Li Y, McIntryre L, Saxena M, Schortgen F, Watts NR, Myburgh J; Fluid-TRIPS and Fluidos Investigators; George Institute for Global Health, The ANZICS Clinical Trials Group, BRICNet, and the REVA research Network. Patterns of intravenous fluid resuscitation use in adult intensive care patients between 2007 and 2014: An international cross-sectional study. PLoS One. 2017 May 12;12(5):e0176292. doi: 10.1371/journal.pone.0176292. eCollection 2017. PMID 28498856